CLINICAL TRIAL: NCT07118891
Title: A First-in-Human Phase 1/2 Study of ABCL635 in Healthy Participants and in Postmenopausal Women With Moderate-to-Severe Vasomotor Symptoms
Brief Title: Study Evaluating ABCL635 for Vasomotor Symptoms of Menopause
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AbCellera Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ABCL635-101; 297103 (Other: Health Canada CTA control number)
Record Dates: First submitted 2025-07-16; First posted 2025-08-12 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-07

CONDITIONS: Vasomotor Symptoms Associated With Menopause; Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- ABCL635 Part A (Experimental): Part A: healthy male and female participants will receive a single dose of ABCL635 administered by subcutaneous (SC) injection
  Interventions: Biological: ABCL635
- Placebo Part A (Placebo Comparator): Part A: Healthy male and female participants will receive a single dose of placebo (dextrose 5% solution) administered by SC injection
  Interventions: Biological: Placebo
- ABCL635 Part B (Experimental): Part B: healthy postmenopausal women with or without VMS will receive up to 3 doses of ABCL635 administered by SC injection
  Interventions: Biological: ABCL635
- Placebo Part B (Placebo Comparator): Part B: healthy postmenopausal women with or without VMS will receive up to 3 doses of placebo (dextrose 5% solution) administered by SC injection
  Interventions: Biological: Placebo
- ABCL635 Part C (Experimental): Part C: postmenopausal women with moderate to severe VMS will receive a single dose of of ABCL635 administered by SC injection
  Interventions: Biological: ABCL635
- Placebo Part C (Placebo Comparator): Part C: postmenopausal women with moderate to severe VMS will receive a single dose o of placebo (dextrose 5% solution) administered by SC injection
  Interventions: Biological: Placebo
- ABCL635 Part C OLE (Experimental): Part C open label extension (OLE): postmenopausal women with moderate to severe VMS who received placebo will receive a single dose of ABCL635 administered by SC injection upon completion of 12-week assessment.
  Interventions: Biological: ABCL635

INTERVENTIONS:
Biological: ABCL635 — Participants will receive SC administrations of ABCL635
  Arms: ABCL635 Part A; ABCL635 Part B; ABCL635 Part C; ABCL635 Part C OLE
Biological: Placebo — Participants will receive SC administration of placebo (5% dextrose solution)
  Arms: Placebo Part A; Placebo Part B; Placebo Part C

SUMMARY:
The purpose of this study is to evaluate the effects of single and multiple doses of ABCL635 administered by subcutaneous (SC) injection to healthy men and to postmenopausal women with or without any vasomotor symptoms (VMS) or hot flashes, and to postmenopausal women with moderate-to-severe VMS associated with menopause. The safety, tolerability, pharmacokinetic (PK) and pharmacodynamic (PD) parameters of ABCL635 will be assessed in all study participants; the effects on frequency and severity of VMS will be assessed in postmenopausal women who experience moderate-to-severe symptoms.

DETAILED DESCRIPTION:
The study consists of 3 parts. In Part A, single ascending doses (SAD) of ABCL635 or placebo will be administered to healthy male and female participants. In Part B, up to 3 multiple ascending doses (MAD) of ABCL635 or placebo will be administered to healthy postmenopausal women with or without VMS. In Part C, a single dose of ABCL635 or placebo will be administered to postmenopausal women experiencing moderate-to-severe VMS associated with menopause. Part C participants receiving placebo will be offered to participate in an open label extension (OLE) cohort and receive a single dose of ABCL635 upon completion of a 12-week assessment.

ELIGIBILITY:
Inclusion Criteria:

* Good general health as determined through a review of their medical history and after conducting a general physical examination
* Body weight ≥ 45 to ≤ 120 kg
* Body mass index (BMI) between 18.5 kg/m2 and 35.0 kg/m2
* Non- or ex-smoker (an ex-smoker is defined as someone who completely stopped using nicotine products for at least 90 days prior to the first study drug administration)
* Healthy man or a postmenopausal woman who is ≥ 40 and ≤ 65 years of age OR a postmenopausal woman with or without VMS and who is ≥ 40 and ≤ 65 years of age OR a postmenopausal woman who is ≥ 40 and ≤ 65 years of age seeking treatment for relief for VMS
* If a woman:

  1. has been compliant with local and/or national guidelines for breast cancer screening with documentation of a mammogram with normal/negative or no clinically significant findings. A screening mammogram may be conducted during study screening period, if needed
  2. has spontaneous amenorrhea for at least 12 consecutive months; or spontaneous amenorrhea for at least 6 months with biochemical criteria of menopause (follicle-stimulating hormone [FSH] > 40 IU/L); or had a bilateral oophorectomy > 6 weeks prior to screening
* If a man:

  1. possess a testosterone concentration of ≥ 15 nmol/L at the time of screening
  2. can procreate and agree to use one of the acceptable contraceptive regimens and not to donate sperm from the first study drug administration to at least 90 days after the last drug administration OR is unable to procreate; defined as surgically sterile

Exclusion Criteria:

* Pregnancy and/or lactation.
* History of abnormal uterine bleeding or endometrial hyperplasia.
* Previous or current history of a malignant tumor, except for basal cell carcinoma.
* Seated pulse rate less than 50 beats per minute (bpm) or more than 100 bpm or a seated blood pressure < 90/50 mmHg or > 140/90 mmHg
* eGFR < 60 mL/min/1.73 m2
* Severe hypersensitivity reactions (like angioedema) to any drugs.
* Significant uncontrolled cardiovascular, pulmonary, gastrointestinal, hepatic, renal, hematologic, neurological, psychiatric, endocrine, immunologic, or dermatologic disease.
* Clinically significant ECG abnormalities
* Syncope or unexplained dizziness.
* Use of any medication (hormonal, prescription, over the counter, herbal, or natural) for the treatment of hot flashes or over-the-counter products (including supplements) containing testosterone less than 28 days prior to study drug administration

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events (AE) | Day 0 to day 197
Number of participants with abnormalities in 12-lead safety electrocardiograms (ECG) | Day 0 to day 197
Number of participants with abnormalities in physical examination | Day 0 to day 197
Number of participants with abnormalities in laboratory parameters, including general biochemistry, hematology, endocrinology, and urinalysis | Day 0 to day 197

SECONDARY OUTCOMES:
Plasma concentrations of ABCL635 | Day 0 to day 197
Incidence of anti-ABCL635 antibodies | Day 0 to day 197
PK parameters; maximum plasma concentration (Cmax) | Day 0 to day 197
PK parameters; time to maximum plasma concentration (Tmax) | Day 0 to day 197
PK parameters; area under the plasma concentration-time curve from zero to the time of the last quantifiable concentration (AUC0-T) | Day 0 to day 197
PK parameters; area under the plasma concentration-time curve from zero to hour 672 (AUC0-672) | Day 0 to day 197
PK parameters; area under the plasma concentration-time curve from zero to infinity (AUC0-∞) | Day 0 to day 197
PK parameters; percent of AUC obtained by extrapolation (%AUCextrap) | Day 0 to day 197
PK parameters; terminal rate constant (λz) | Day 0 to day 197
PK parameters; apparent plasma clearance of drug after extravascular administration (CL/F) | Day 0 to day 197
PK parameters; apparent volume of distribution after extravascular administration (Vz/F) | Day 0 to day 197
PK parameters; half-life (Thalf) | Day 0 to day 197

OTHER OUTCOMES:
Mean change from baseline to each study week in the frequency of moderate and severe VMS (VMSM-S frequency) | up to day 141 (Part C)
Mean change from baseline to each study week in the severity of moderate and severe VMS (VMSM-S severity) | up to day 141 (Part C)
Mean change from baseline to each study week in the frequency of all reported VMS (VMSTotal frequency). | up to day 141 (Part C)
Mean change from baseline to each study week in the moderate to severe hot flash score (HFM-S). | up to day 141 (Part C)
  The moderate to severe hot flash score (HFM-S) is a metric that combines the frequency and severity of hot flashes:
  * The daily score is calculated as follows: (number of moderate hot flashes x 2) + (number of severe hot flashes x 3)
  * The weekly score is the average daily score over seven days. A negative change in the score from Baseline to Week 1 indicates a reduction in the severity and frequency of hot flashes
Mean change from baseline to each study week in the total hot flash score (HFTotal). | up to day 141 (Part C)
  he total hot flash score (HFTotal) is a metric that combines the frequency and severity of hot flashes:
  * The daily score is calculated as follows: (number of mild hot flashes x 1) + (number of moderate hot flashes x 2) + (number of severe hot flashes x 3)
  * The weekly score is the average daily score over seven days. A negative change in the score from Baseline to Week 1 indicates a reduction in the severity and frequency of hot flashes.
Mean change in the Menopause-Specific Quality of Life Questionnaire (MENQOL) 4-domain scores (ie, physical, vasomotor, psychosocial, and sexual) from baseline to weeks 1, 2, 3, 4, 5, 9, and 13 | up to day 141 (Part C)
  The Mean change in the Menopause-Specific Quality of Life Questionnaire (MENQOL) measures the impact of menopause symptoms over the last week.
  The questionnaire has 29 items across four domains: vasomotor (items 1 to 3), psychosocial (items 4 to 10), physical (items 11 to 26), and sexual (items 27 to 29). Items pertaining to a specific symptom are rated as present or not present, and if present, how bothersome on a 0 (not bothersome) to 6 (extremely bothersome) scale.
  The mean change in the MENQOL domain scores will be assessed from Baseline to each week measured. A negative change in the score from Baseline to each week measured indicates an improvement in quality of life.
Mean change in the Patient-Reported Outcomes Measurement Information System Sleep Disturbance 8b Short Form (PROMIS-SD-SF-8b) total score from baseline to weeks 1, 2, 3, 4, 5, 9, and 13. | up to day 141 (Part C)
  The PROMIS-SD-SF-8b assesses the perception of sleep quality, sleep depth, and any perceived difficulties related to getting and staying asleep. Questions are scored using the following scale: 1 (very much), 2 (quite a bit), 3 (somewhat), 4 (a little bit), and 5 (not at all).
  The mean change in the PROMIS-SD-SF-8b score will be assessed from Baseline to each week measured. A positive change in the score from Baseline to each week measured indicates a reduction in sleep disturbance.
Frequency of Patient Global Impression of Change in VMS (PGI-C VMS) responses at weeks 2, 3, 4, 5, 9, and 13. | up to day 141 (Part C)
  The Patient Global Impression of Change (PGI-C) for vasomotor symptoms (VMS) rates the perception of their hot flashes and night sweats at each designated timepoint compared to the start of the study. The response is a seven-point scale ranging from "much better" to "much worse." The frequency of each PGI-C VMS score will be reported at each scheduled timepoint.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, Principal Investigator — Altasciences Company Inc.
Locations (7):
- Canada (7):
  - Mount Saint Joseph Hospital Clinical Trials Phase 1 Unit, Vancouver, British Columbia
  - Centricity Research, Toronto, Ontario
  - Altasciences Company Inc., Mount Royal, Quebec
  - Clinique RSF Inc., Québec, Quebec
  - Diex Recherche Sherbrooke, Sherbrooke, Quebec
  - Diex Recherche Trois-Rivières, Trois-Rivières, Quebec
  - Diex Recherche Victoriaville, Victoriaville, Quebec

IPD SHARING:
Plan to Share IPD: No